CLINICAL TRIAL: NCT02823002
Title: The Impact of Anesthetic Injection Rate, Temperature and Buffering on Pain Perception During Dermatologic Procedures: a Multicenter, Single-blinded Randomized Control Trial
Brief Title: Pain Perception: Lidocaine Rate/Temp/Buffer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Murad Alam, Professor in Dermatology, Otolaryngology-Head and Neck Surgery, and Surgery, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: STU00202894
Record Dates: First submitted 2016-06-27; First posted 2016-07-06 (Estimated); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Ampholyte Mixtures; Lidocaine; Buffers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Slow, Room Temperature (Experimental): In Part A, subject will be randomized to receive an injection of lidocaine that is slow at room temperature, rapid at room temperature, slow at warm temperature, or rapid at warm temperature.
  Interventions: Procedure: Slow, Room Temperature Injection; Drug: Lidocaine; Drug: Buffer
- Rapid, Room Temperature (Experimental): In Part A, subject will be randomized to receive an injection of lidocaine that is slow at room temperature, rapid at room temperature, slow at warm temperature, or rapid at warm temperature.
  Interventions: Procedure: Rapid, Room Temperature Injection; Drug: Lidocaine; Drug: Buffer
- Slow, Warmed (Experimental): In Part A, subject will be randomized to receive an injection of lidocaine that is slow at room temperature, rapid at room temperature, slow at warm temperature, or rapid at warm temperature.
  Interventions: Procedure: Slow, Warm Temperature Injection; Drug: Lidocaine; Drug: Buffer
- Rapid, Warmed (Experimental): In Part A, subject will be randomized to receive an injection of lidocaine that is slow at room temperature, rapid at room temperature, slow at warm temperature, or rapid at warm temperature.
  Interventions: Procedure: Rapid, Warm Temperature Injection; Drug: Lidocaine; Drug: Buffer
- Buffered (Experimental): In Part B, subject will be randomized to receive an injection of lidocaine that is buffered or non-buffered.
  Interventions: Procedure: Buffered Injection; Drug: Lidocaine; Drug: Buffer
- Non-Buffered (Placebo Comparator): In Part B, subject will be randomized to receive an injection of lidocaine that is buffered or non-buffered.
  Interventions: Procedure: Non-Buffered Injection; Drug: Lidocaine

INTERVENTIONS:
Procedure: Slow, Room Temperature Injection — The room temperature local anesthetic agent will be administered by slow infiltration.
  Arms: Slow, Room Temperature
Procedure: Rapid, Room Temperature Injection — The room temperature local anesthetic agent will be administered by rapid infiltration.
  Arms: Rapid, Room Temperature
Procedure: Slow, Warm Temperature Injection — The warmed local anesthetic agent will be administered by slow infiltration.
  Arms: Slow, Warmed
Procedure: Rapid, Warm Temperature Injection — The warmed local anesthetic agent will be administered by rapid infiltration.
  Arms: Rapid, Warmed
Procedure: Buffered Injection — One side of the body will be randomized to receive an injection of the buffered agent, while the contralateral side will be assigned to receive an injection of the unbuffered anesthetic agent.
  Arms: Buffered
Procedure: Non-Buffered Injection — One side of the body will be randomized to receive an injection of the buffered agent, while the contralateral side will be assigned to receive an injection of the unbuffered anesthetic agent.
  Arms: Non-Buffered
Drug: Lidocaine — Injectable lidocaine solution (Lidocaine Hydrochloride and Epinephrine)
Drug: Buffer — Sodium Bicarbonate
  Arms: Buffered; Rapid, Room Temperature; Rapid, Warmed; Slow, Room Temperature; Slow, Warmed

SUMMARY:
This study will collect data from multiple academic institutions. The primary objective for part A of this study is to determine the impact of anesthetic injection rate and temperature on pain perception during dermatologic procedures, and the objective for the part B of this study is to determine if buffering of the anesthetic solution alters pain perception.

This study is a pilot study designed to determine feasibility of these procedures.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are undergoing dermatologic procedures.
* Subjects ages 18-89 year old.
* The subjects have the willingness and the ability to understand and provide informed consent and communicate with the investigator.

Exclusion Criteria:

* Subjects who are allergic to lidocaine.
* History of bleeding tendency or coagulopathy.
* Pregnant or lactating.
* Active skin disease or skin infection in the treatment area.
* Unable to understand the protocol or give informed consent.
* Any other condition, in the professional opinion of the investigator, that would potentially affect response or participation in the clinical study, or would pose as an unacceptable risk to the subject.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2016-06; Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Pain on a Visual Analog Scale (VAS) | intraoperative
  Subjects will rate the pain VAS score immediately after the needle is withdrawn. They will be asked to rate the pain of the injection of the solution. VAS pain scale is rated on a 10 cm scale with 0 cm being no pain and 10 cm being extremely painful.

CONTACTS AND LOCATIONS:
Overall Officials: Murad Alam, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University Department of Dermatology, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided